CLINICAL TRIAL: NCT01700725
Title: Nasal Irrigation for Chronic Rhinosinusitis and Fatigue in Patients With Gulf War Illness
Brief Title: Gulf War Illness Nasal Irrigation Study
Acronym: GWINIS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GW100054 US Dept of Defense; 2011-0843 (Other: HS IRB)
Record Dates: First submitted 2012-08-14; First posted 2012-10-04 (Estimated); Results first posted 2019-05-21 (Actual); Last update posted 2019-05-21 (Actual); Status verified 2019-05

CONDITIONS: Persian Gulf Syndrome; Chronic Sinusitis; Fatigue; Acute Sinusitis
Keywords: Gulf War Illness; xylitol; nasal irrigation; Desert Storm; Persian Gulf Conflicts; neti pot; cytokines; nasal mucus; inflammatory mediator; lactoferrin; lysozyme
MeSH Terms: conditions — Persian Gulf Syndrome; Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Nasal Irrigation - Saline (Experimental): nasal irrigation using saline plus routine care for symptoms of CRS and fatigue
  Interventions: Other: Nasal Irrigation - Saline
- Nasal Irrigation - Xylitol (Experimental): Nasal Irrigation with Xylitol plus routine care for symptoms of CRS and fatigue
  Interventions: Drug: Nasal Irrigation - Xylitol
- Control Group (No Intervention): Control group subjects continue to use routine care only

INTERVENTIONS:
Other: Nasal Irrigation - Saline — Liquid-based nasal irrigation (NI) is performed using a nasal irrigation cup ("neti pot"), a simple hand-held vessel that uses the force of gravity to gently irrigate the user's nasal cavity. Subjects will be requested to perform NI twice daily. The subjects will prepare the saline solution by themselves using the study-provided kit which will include packets of salt powder and the neti pot; subjects will dissolve the powder in lukewarm tap water to achieve a 2% buffered saline solution. The solution is then delivered to the nasal cavity using neti pot.
  Other Names: 2% buffered saline
  Arms: Nasal Irrigation - Saline
Drug: Nasal Irrigation - Xylitol — Liquid-based nasal irrigation (NI) is performed using a nasal irrigation cup ("neti pot"), a simple hand-held vessel that uses the force of gravity to gently irrigate the user's nasal cavity. Subjects will be requested to perform NI twice daily. The subjects will prepare the Xylitol solution by themselves using the study-provided kit which will include packets of Xylitol powder and the neti pot; subjects will dissolve the powder in lukewarm tap water to achieve a 5% Xylitol solution. The solution is then delivered to the nasal cavity using neti pot.
  Other Names: 5% Xylitol solution
  Arms: Nasal Irrigation - Xylitol

SUMMARY:
The purpose of this study is to determine whether nasal irrigation with Xylitol or saline are effective in the treatment of chronic rhinosinusitis and fatigue symptoms associated with Gulf War Illness.

DETAILED DESCRIPTION:
Background: Gulf War Illness (GWI) results in tremendous impact to quality of life. Symptoms of chronic rhinosinusitis (CRS) and fatigue are the first (47%) and third (41%) most common symptoms of patients with GWI, respectively. These symptoms are biologically characterized by a milieu of elevated levels of proinflammatory cytokines; to date, the profile of these cytokines in serum and nasal secretions is incompletely understood and has not been assessed in response to therapy. Nasal irrigation (NI) is a therapy which bathes the nasal cavity with a solution (liquid). There are two promising forms of NI; saline NI (S-NI) is hypothesized to improve sinus symptoms by thinning and clearing mucus and inflammatory mediators, decreasing mucosal edema and improving ciliary function. Xylitol NI (X-NI) has been shown to change the salinity of the mucosal surface resulting in enhanced antimicrobial properties. Although NI is an evidence-based adjunctive therapy for CRS and has been reported to be effective for CRS and fatigue, it has not been assessed in a GWI population.

Specific Aims, Hypotheses and Study Design: The specific aims of this proposal are to determine whether routine care plus S-NI, or X-NI, compared to routine care alone, result in improved health-related quality of life (HRQoL), are cost-effective and decrease proinflammatory bias in subjects with GWI who suffer from CRS and fatigue.

Consistent with our specific aims, we will test the following hypotheses: In an RCT setting, at 26 weeks post-enrollment, adults with GWI and symptoms of CRI and fatigue, treated with routine care plus S-NI or X-NI, compared to those treated with routine care alone, will demonstrate:

H1: improved HRQoL: a) sinus-disease specific HRQoL as evaluated by the validated Sinonasal Outcomes Test (SNOT-20) questionnaire (primary outcome measure); b) fatigue-specific HRQoL as assessed by the validated questionnaire, the Multidimensional Fatigue Inventory (MFI); and c) overall HRQoL as assessed by the validated questionnaire the Medical Outcomes Survey Short Form-36 (SF-36; mental and physical health domains) augmented with 18 sleep- and breathing related questions.

H.2: greater cost-effectiveness as measured by the average cost of the intervention divided by the average effectiveness (as assessed by a improvement in SNOT-20 scores), and reported as the "dollars spent per subject restored to health."

H.3: improved treatment satisfaction as assessed by a single-item treatment satisfaction score and a qualitative exit interview.

H.4: improved proinflammatory bias: a) reduced activation and dysregulation of proinflammatory pathways as determined by a reduction in URI-specific inflammatory cytokines in serum and nasal secretions; and b) improved serum-based complete blood count, sedimentation rate or C-reactive protein, or nasal swab-based neutrophil or eosinophil counts.

Study Design: 26 week duration of follow-up, 3-arm RCT (N=75). All groups will utilize routine care for their GWI and symptoms of CRS and fatigue. Groups 1 and 2 will in addition add S-NI or X-NI twice daily to their routine care, respectively. Group 3 will continue to use routine care with no other additions (control group); control group participants will be offered NI training and related materials (xylitol or saline per subject preference) after they complete their 26-week follow-up period.

Impact: Positive findings would suggest a number of important effects:

* Statistically positive results on HRQoL outcome measures would suggest that NI can provide effective adjunctive therapy for CRS and fatigue in adults with GWI, improving health of affected patients and potentially providing gains to society through reduced health care utilization and absenteeism related costs.
* Positive biomarker findings would contribute to our better understanding of the etiology of CRS and fatigue in the GWI population and of possible biological pathways underlying the NI efficacy.
* The finding that either form of NI is cost effective would provide economic justification for its clinical use.

ELIGIBILITY:
Inclusion Criteria:

* English fluency and basic reading and writing literacy.
* Deployment to the Persian Gulf (e.g., Iraq, Kuwait, Saudi Arabia) for the purpose of Operation Desert Shield or Operation Desert Storm during the first Gulf War (1990-1991).
* Meeting criteria for a diagnosis of GWI as based on the "Kansas" GWI case definition; only the Kansas case definition (from among the several currently used case definitions) can differentiate between Gulf War-deployed and non-deployed Gulf era veterans.
* Meeting criteria for a diagnosis of chronic rhinosinusitis (CRS) using self-reported symptoms and based on clinical guidelines; eligible subjects will report: • sinonasal symptoms for at least 12 weeks; • a constellation of sinonasal symptoms including either two or more major factors, or 1 major and 2 minor factors (see Table 1 below), or chronic nasal purulence for 12 or more weeks; and • a moderate to severe HRQoL impact (≥ 3 points on a 0-10 Likert severity scale) as assessed by a single item question:11 "What has been the average level of your sinus symptoms daily over the past month on a 0-10 scale?" This item is consistent with eligibility criteria used in prior NI studies.
* Chronic fatigue of moderate-to-severe severity defined as scoring at least 3 points on a single question (0-10 Likert scale): "What has been the average level of your daily fatigue over the past month on a 0-10 scale?"

Exclusion Criteria:

* Self-reported pregnancy.
* Current use of liquid NI or xylitol nasal spray; regular use is defined as 1 or more irrigations weekly for 3 consecutive weeks.
* Self-reported neurological or musculoskeletal conditions that could facilitate aspiration, or patients who otherwise cannot physically perform the NI procedure.
* Self-reported borderline personality disorder.
* Inability or stated reluctance to reliably participate in study activities.
* Severe or unstable mental health problems that would preclude safe or reliable study participation as based on an in-person evaluation by a psychiatry team; active delusional disorder, depressive disorder or alcohol/drug abuse or dependence will be a primary target of this interview using both a structured clinical interview (MINI ref) and psychiatry team evaluation.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Molander, MD, Principal Investigator — US Department of Veterans Affairs, William S. Middleton Memorial Veterans Hospital; David P Rabago, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin General Clinical Research Center, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Hayer SD, Rabago DP, Amaza IP, Kille T, Coe CL, Zgierska A, Zakletskaia L, Mundt MP, Krahn D, Obasi CN, Molander RC. Effectiveness of nasal irrigation for chronic rhinosinusitis and fatigue in patients with Gulf War illness: protocol for a randomized controlled trial. Contemp Clin Trials. 2015 Mar;41:219-26. doi: 10.1016/j.cct.2015.01.008. Epub 2015 Jan 24. PMID 25625809

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nasal Irrigation - Xylitol | Nasal Irrigation - Saline | Control Group
Started | 14 | 14 | 12
Completed | 14 | 14 | 12
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nasal Irrigation - Xylitol | Nasal Irrigation - Saline | Control Group | Total
Number analyzed (Participants) | 14 | 14 | 12 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (9.2) | 52.7 (6.7) | 55.0 (7.7) | 53.8 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 3 | 8
  Male | 10 | 13 | 9 | 32
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 12 | 8 | 11 | 31
  White Hispanic | 1 | 2 | 1 | 4
  African American | 1 | 1 | 0 | 2
  Asian | 0 | 1 | 0 | 1
  Pacific Islander / Hawaiian | 0 | 1 | 0 | 1
  Multiple Races | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 14 | 14 | 12 | 40
Education [Count of Participants; unit: Participants]
  Highschool or Less | 1 | 1 | 1 | 3
  Some College | 8 | 8 | 4 | 20
  College Graduate | 5 | 5 | 7 | 17
Sinusitis Symptoms [Mean (Standard Deviation); unit: years] | 20.5 (7.8) | 16.4 (9.9) | 22.4 (2.3) | 19.8 (7.7)
Fatigue [Mean (Standard Deviation); unit: years] | 19.3 (8.4) | 19.9 (6.0) | 23.8 (3.1) | 20.7 (6.6)
SNOT-20 [Mean (Standard Deviation); unit: units on a scale] — Sinus disease specific quality of life will be measured using the total score of this validated 20 item questionnaire. It is a reliable and valid outcome measure for patients with CRS (Cronbach's α 0.9, test-retest r = 0.9) that describes the health burden and is sensitive to clinical change. Patients who are more affected by CRS tend to have greater SNOT-20 scores (P < 0.01). The SNOT-20 score is expected to improve in NI-treated subjects compared to controls.The total range of possible scores is 0-100. The higher the score, the worse the symptoms.
  units on a scale | 50.8 (14.7) | 47.6 (13.7) | 47.2 (8.7) | 48.5 (12.7)
SF-36 [Mean (Standard Deviation); unit: units on a scale] — SF-36 is a validated questionnaire designed to assess health status, function and overall health related quality of life. It includes one multi-item scale assessing 8 areas: 1) limitations in physical activities; 2) limitations in social activities; 3) limitations in usual role activities (physical problems); 4) bodily pain; 5) general mental health; 6) limitations in usual role activities (emotional problems); 7) vitality; and 8) general health perceptions. Eighteen relevant sleep and breathing related questions to the SF-36. The total range is 0-100. The lower the score, the more disability.
  units on a scale | 51.1 (15.8) | 59.0 (17.6) | 62.7 (14.1) | 57.3 (16.3)
MFI [Mean (Standard Deviation); unit: units on a scale] — The Multidimensional Fatigue Inventory is a validated disease specific outcome measure for fatigue. The instrument has good internal consistency (average Cronbach's alpha 0.84). Fatigue is expected to improve in the NI-treated patients compared to controls. The total range of possible scores is 0-100. The higher the score, the more fatigue.
  units on a scale | 59.4 (5.4) | 60.5 (6.0) | 61.7 (4.7) | 60.4 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Sino-Nasal Outcome Test (SNOT-20) Score From Baseline
Description: Sino-Nasal Outcome Test (SNOT-20) is a recommended tool for clinical trial research involving CRS. Sinus disease specific quality of life will be measured using the total score of this validated 20 item questionnaire. It is a reliable and valid outcome measure for patients with CRS (Cronbach's α 0.9, test-retest r = 0.9) that describes the health burden and is sensitive to clinical change. Patients who are more affected by CRS tend to have greater SNOT-20 scores (P < 0.01). The SNOT-20 score is expected to improve in NI-treated subjects compared to controls. Findings of the PI's prior RCT of adults with CRS are consistent with the above evidence. The total range of possible scores is 0-100. The higher the score, the worse the symptoms.
Time Frame: Change from baseline week 8, change from baseline week 26
Population: Data from one participant in the control group and two participants in the Saline group at 26 weeks was unable to be collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nasal Irrigation - Xylitol | Nasal Irrigation - Saline | Control Group
Number analyzed (Participants) | 14 | 14 | 12
score on a scale
  Baseline to Week 8 | -16.9 (4.9) | -8.8 (5.0) | -3.4 (5.3)
  Baseline to Week 26: number analyzed (Participants) | 14 | 12 | 11
  Baseline to Week 26 | -18.9 (4.9) | -16.9 (5.3) | -3.5 (5.6)

2. Secondary Outcome: Change in Multidimensional Fatigue Inventory (MFI) Over Baseline
Description: The Multidimensional Fatigue Inventory is a validated disease specific outcome measure for fatigue. The instrument has good internal consistency (average Cronbach's alpha 0.84). Construct validity was established after comparisons between and within groups, assuming differences in fatigue based on differences in circumstances and/or activity level. Convergent validity was investigated by correlating the MFI-scales with a Visual Analogue Scale measuring fatigue. Fatigue is expected to improve in the NI-treated patients compared to controls. The total range of possible scores is 0-100. The higher the score, the more fatigue.
Time Frame: Baseline to weeks 8 & 26
Population: Data from several participants was unable to be collected at various timepoints.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nasal Irrigation - Xylitol | Nasal Irrigation - Saline | Control Group
Number analyzed (Participants) | 12 | 14 | 12
score on a scale
  Baseline to Week 8 | 0.6 (2.4) | 0.9 (2.3) | 0.5 (2.5)
  Baseline to Week 26: number analyzed (Participants) | 12 | 12 | 8
  Baseline to Week 26 | 1.9 (2.8) | -1.4 (2.4) | 10.4 (3.0)

3. Secondary Outcome: Change in Medical Outcomes Survey Short Form-36 (SF-36) Over Baseline
Description: SF-36 is a validated questionnaire designed to assess health status, function and overall health related quality of life. The SF-36 includes one multi-item scale that assesses eight health concepts: 1) limitations in physical activities because of health problems; 2) limitations in social activities because of physical or emotional problems; 3) limitations in usual role activities because of physical health problems; 4) bodily pain; 5) general mental health (psychological distress and well-being); 6) limitations in usual role activities because of emotional problems; 7) vitality (energy and fatigue); and 8) general health perceptions. Gulf War Illness and chronic rhinosinusitis both affect sleep and breathing parameters. Prior studies suggest that both may be improved with SNI in some subjects. Eighteen relevant sleep and breathing related questions to the SF-36. The total range is 0-100. The lower the score, the more disability.
Time Frame: Baseline and weeks 8 & 26
Population: Data from one participant at 26 weeks in the control group was unable to be collected.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Nasal Irrigation - Xylitol | Nasal Irrigation - Saline | Control Group
Number analyzed (Participants) | 14 | 14 | 12
score on a scale
  Baseline to Week 8 | 1.1 (3.5) | 3.9 (3.6) | -0.1 (3.8)
  Baseline to Week 26: number analyzed (Participants) | 14 | 14 | 11
  Baseline to Week 26 | 6.4 (3.5) | 7.3 (3.6) | 2.0 (4.0)

ADVERSE EVENTS:
Time Frame: Up to 26 weeks
Arm/Group | Nasal Irrigation - Xylitol | Nasal Irrigation - Saline | Control Group
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/12
Other Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes